CLINICAL TRIAL: NCT05882318
Title: Evaluating Effectiveness of Sensory and Subsensory Stimulation Amplitudes With eCoin® Tibial Nerve Stimulation in Urgency Urinary InContinence Episodes and Quality of Life
Brief Title: Effectiveness of eCoin at Sensory and Subsensory Amplitudes
Acronym: ESSENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valencia Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-6133
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Urge Incontinence
Keywords: Neuromodulation; eCoin device; Stimulation; Tibial nerve
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sensory (Experimental): Participants in the sensory treatment arm will be programmed to their sensory threshold.
  Interventions: Device: eCoin Peripheral Neurostimulator System
- Subsensory (Experimental): Participants in the subsensory treatment arm will be programmed to approximately 75% of their sensory threshold.
  Interventions: Device: eCoin Peripheral Neurostimulator System

INTERVENTIONS:
Device: eCoin Peripheral Neurostimulator System — The eCoin device is a leadless, coin-sized tibial neurostimulator for treatment of urgency urinary incontinence. It emits a dome-shaped electrical field to deliver low-duty cycle stimulation to the tibial nerve. The device is to be implanted under local anesthetic in the lower leg, and once activated delivers automatic 30-minute treatment sessions without the need for patient management.

SUMMARY:
The goal of this prospective, multi-center, double-blinded randomized controlled is to learn about effectiveness and QOL with eCoin at two different amplitude settings in subjects with urge urinary incontincence (UUI). The main question it aims to answer is:

* The reduction in UUI episodes per day on a 3-day voiding diary in both groups after 3 months of therapy

Participants will be implanted with the eCoin device and randomized to either a sensory or subsensory stimulation group and complete voiding diaries and patient reported-outcomes through 3 months of therapy. After 3 months, subjects will be unblinded and reprogramming will be offered. Subjects will be followed for an additional month to a total of 4 months.

ELIGIBILITY:
Key Inclusion Criteria:

1. Individual with diagnosis of overactive bladder with urgency urinary incontinence - daily UUI with a predominantly urgency component
2. Individual is intolerant of or has an inadequate response to any of anticholinergics, β3-adrenoceptor agonists, onabotulinumtoxinA, or who have undergone percutaneous tibial nerve stimulation (PTNS).
3. Individual is determined to be a suitable surgical candidate by physician.

Key Exclusion Criteria:

1. Individual is not appropriate for eCoin therapy based upon the US FDA-approved IFU requirements.
2. Individual has predominantly stress urinary incontinence (greater than 1/3 of leaks on baseline diary are stress).
3. Individual has clinically significant bladder outlet obstruction.
4. Individual has an active urinary tract infection at time of enrollment or has had four or more symptomatic UTI's in the last 12 months.
5. Individual has significant lower urinary tract pain or has been diagnosed with interstitial cystitis or bladder pain syndrome that is actively being managed.
6. Individual has post void residual greater than 200 cc.
7. Individual has an active diagnosis of bladder, urethral, or prostate cancer.
8. Individual has had a prior anti-stress incontinence surgery within the last year.
9. Individual has uncontrolled diabetes mellitus (Hemoglobin A1C>7).
10. Individual is neutropenic or immune-compromised.
11. Individual has lower extremity pathology such as:

    1. Previous surgery and/or significant scarring at the planned implant location
    2. Ongoing dermatologic condition at the implant site, including but not limited to dermatitis and autoimmune disorders
    3. Clinically significant peripheral neuropathy in the lower extremities
    4. Pitting edema at the implant location (≥ 2+ is excluded)
    5. Inadequate skin integrity or any evidence of an infection or inflammation in either lower leg
    6. Moderate to severe varicose veins
    7. Open wounds or recent trauma
    8. Arterial and/or vasculitis disease in the lower extremities
    9. Chronic venous insufficiency with a history of skin change (hyperpigmentation, lipodermatosclerosis, ulceration) in the ankle region
12. Individual has neurogenic bladder dysfunction.
13. Individual is aware that he or she will need an MRI scan other than a head/neck/shoulder MRI during the study period.
14. Any condition that, in the investigator's opinion, would preclude participation in the study (e.g., comorbidity that places subject at increased risk for surgical intervention, medical condition that may increase the risk associated with study participation or may interfere with interpretation of study results, inability to adhere to the visit schedule, such as morbid obesity, clotting or bleeding disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Genesis Research, Downey, California
  - Urology Associates of Central California, Fresno, California
  - The Iowa Clinic, Ankeny, Iowa
  - Cypress Medical Research Center, Wichita, Kansas
  - Adult & Pediatric Urology P.C., Omaha, Nebraska
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Institute for Female Pelvic Medicine, Allentown, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were excluded from randomization following enrollment. Both were due to withdraw of consent.
Groups:
- Sensory: eCoin Peripheral Neurostimulator System: The eCoin device is a leadless, coin-sized tibial neurostimulator for treatment of urgency urinary incontinence. It emits a dome-shaped electrical field to deliver low-duty cycle stimulation to the tibial nerve. The device is to be implanted under local anesthetic in the lower leg, and once activated delivers automatic 30-minute treatment sessions without the need for patient management.
  Participants in the sensory treatment arm are programmed to their sensory threshold.
- Subsensory: eCoin Peripheral Neurostimulator System: The eCoin device is a leadless, coin-sized tibial neurostimulator for treatment of urgency urinary incontinence. It emits a dome-shaped electrical field to deliver low-duty cycle stimulation to the tibial nerve. The device is to be implanted under local anesthetic in the lower leg, and once activated delivers automatic 30-minute treatment sessions without the need for patient management.
  Participants in the subsensory treatment arm are programmed to approximately 75% of their sensory threshold.
Period: Overall Study
Arm/Group | Sensory | Subsensory
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The number of baseline participants refers to the number of participants who were implanted and randomized into a study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensory | Subsensory | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13) | 65 (14) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 15 | 33
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only the per-protocol population (N=30) was analyzed for baseline demographics.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 17 | 15 | 32
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 30
Smoking Status, Current Smoker [Count of Participants; unit: Participants] | 0 | 0 | 0
Baseline UUI Episodes per Day [Mean (Standard Deviation); unit: UUI Episodes per day] — Population: All available baseline UUI data.
  UUI Episodes per day
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 4.91 (2.12) | 5.9 (3.01) | 5.39 (2.6)
Baseline HRQL Score [Mean (Standard Deviation); unit: HRQL Score] — Patient reported quality of life as assessed by the Health Related Quality of Life (HRQL) portion of the Overactive Bladder questionnaire (OABq) survey
  Higher scores on the HRQL portion indicate better quality of life. The maximum HRQL domain score is 100 (best) and the minimum HRQL score is 0 (worst). Population: All available baseline HRQoL Data
  HRQL Score
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 53.07 (18.67) | 53.13 (22.13) | 53.1 (20.11)

OUTCOME MEASURES:

1. Primary Outcome: Change in UUI Episodes Per Day
Description: The primary endpoint is to explore the effect of two different eCoin amplitude settings on the change of UUI episodes per day on a 3-day voiding diary.
  A negative number shows a reduction in UUI episodes per day which means symptoms have improved since baseline.
  A positive number shows an increase in UUI episodes per day which means symptoms have worsened since baseline.
Time Frame: 3 months post-activation
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: UUI episodes per day
Arm/Group | Sensory | Subsensory
Number analyzed (Participants) | 13 | 17
UUI episodes per day | -2.1 (2.42) | -2.73 (1.8)

2. Secondary Outcome: Change in UUI Episodes Per Day
Description: Change in the number of urgency urinary incontinence episodes per day on a 3-day voiding diary.
  A negative number shows a reduction in UUI episodes which means symptoms have improved since baseline.
  A positive number shows an increase in UUI episodes per day which means symptoms have worsened since baseline.
Time Frame: 2 months post-activation
Population: Per-Protocol Population with available UUI data at 2 months post-activation
Measure: Mean (Standard Deviation); unit: UUI episodes per day
Arm/Group | Sensory | Subsensory
Number analyzed (Participants) | 12 | 17
UUI episodes per day | -2.75 (1.9) | -2.14 (2.58)

3. Secondary Outcome: Change in UUI Episodes Per Day
Description: A secondary endpoint is to explore the change in UUI episodes per day on a 3-day voiding diary.
  A negative number shows a reduction in UUI episodes per day which means symptoms have improved since baseline.
  A positive number shows an increase in UUI episodes per day which means symptoms have worsened since baseline.
Time Frame: 4 months post-activation
Population: Per-Protocol Population with available UUI data at 4 months post-activation
Measure: Mean (Standard Deviation); unit: UUI episodes per day
Arm/Group | Sensory | Subsensory
Number analyzed (Participants) | 13 | 17
UUI episodes per day | -2.59 (2.6) | -2.96 (2.12)

4. Secondary Outcome: Change in Overactive Bladder Health Related Quality of Life (HRQL)
Description: Change from baseline in the patient reported quality of life as assessed by the Health Related Quality of Life (HRQL) portion of the Overactive Bladder questionnaire (OABq) survey.
  Higher scores on the HRQL portion indicate better quality of life. The maximum HRQL domain score is 100 (best) and the minimum HRQL score is 0 (worst).
  A positive change in score indicates an improvement in quality of life.
Time Frame: 2 and 3 months post-activation
Population: Per-Protocol Population all available data
Measure: Mean (Standard Deviation); unit: Change in HRQL Score
Arm/Group | Sensory | Subsensory
Number analyzed (Participants) | 13 | 17
Change in HRQL Score
  2 months: number analyzed (Participants) | 12 | 17
  2 months | 25.87 (21.6) | 22.78 (24.19)
  3-months | 18.15 (22.63) | 22.59 (24.95)

5. Secondary Outcome: Change in Overactive Bladder Health Related Quality of Life (HRQL)
Description: Change from baseline in patient reported quality of life as assessed by the Health Related Quality of Life (HRQL) portion of the Overactive Bladder questionnaire (OABq) survey.
  Higher scores on the HRQL indicate better quality of life. The maximum HRQL domain score is 100 (best) and the minimum HRQL score is 0 (worst).
  A positive change in score indicates an improvement in quality of life.
Time Frame: 4 months post-activation
Population: Per-Protocol Population with available UUI data at 4 months post-activation
Measure: Mean (Standard Deviation); unit: Change in HRQL Score
Arm/Group | Sensory | Subsensory
Number analyzed (Participants) | 13 | 17
Change in HRQL Score | 22.03 (25.56) | 32.09 (26.2)

ADVERSE EVENTS:
Time Frame: 4 months post-activation
Description: The analysis set is comprised of "treatment emergent" adverse events, defined as device- or procedure-related adverse events occurring on or after implantation or attempted implantation of eCoin. Safety results are summarized for all implanted patients. At each follow-up visit, adverse events were recorded on the CRF. Patients were unblinded following the 3 month visit and had the option to reprogram their devices. Results are reported based on the patient's original treatment arm.
Arm/Group | Sensory | Subsensory
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 7/18 | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensory (N=18) | Subsensory (N=18)
Medical Device Site Erythema (General disorders) | 0 (0) | 1 (1)
Post Procedural Discomfort (General disorders) | 0 (0) | 1 (1)
Incision Site Impaired Healing (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision Site Discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Implant Site Oedema (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Cellulitis, Medical Device Site Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Pain, Implant Site Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Site Incision Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision Site Pain, Incision Site Hyperaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Device Stimulation issue (Product Issues) | 1 (1) | 0 (0)
Dermatitis Contact (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Implant Site Ulcer (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Implant Site Pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05882318/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT05882318/SAP_001.pdf